CLINICAL TRIAL: NCT03474393
Title: A Randomised Trial of Evaluating a Systematic Intensive Therapy Using Continuous Glucose Monitoring (CGM) and Flash Glucose Monitoring (FGM) in Clinical Diabetes Care
Brief Title: A Evaluation of Systematic Intensive Therapy Using CGM/FGM in Clinical Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIT-CGM/FGM
Record Dates: First submitted 2018-03-01; First posted 2018-03-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-02

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal diabetes care (No Intervention): Continue with their normal diabetes care. Come in for control visits
- Systematic intensive therapy (Experimental): Intensive Internet and telephone contact for 4 months and Control visits
  Interventions: Other: systematic intensive therapy

INTERVENTIONS:
Other: systematic intensive therapy — intensive telephone och internet Contact with diabetes nurse for coaching and guidance over 4 months and 4 Control visits
  Arms: Systematic intensive therapy

SUMMARY:
This study aims to analyse if intensive systematic treatment via internet and telephone during 4 months improved HbA1c for persons with type 1 diabetes which are already treated with CGM or FGM, and if the effect continuous for 1-2 years after the intervention stops. Time in Hypoglycaemia, treatment satisfaction, Diabetes distress and hypoglycaemia fear will even be analysed.

A randomised, non-blinded, multi-centre, clinical study for persons with type 1 diabetes and hbA1c ≥ 58mmol/mol and treated with CGM or FGM.

The control group continuous its normal diabetes care with study visits at randomisation, 10, 18, 32, and 52 weeks for HbA1c and to fill in questionnaires.

The intervention group will have contact with the study team on a weekly basis, when mean blood glucose levels the previous week are elevated. They will receive help with analysing data and advice on how to improve their glucose values. They will even meet the study team at randomisation, 10, 18, 32, and 52 weeks for HbA1c and to fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before trial-related activities (i.e., any activity that would not have been performed during routine patient management)
* Clinical diagnosis of Type 1 diabetes
* Adult patients over 18 years of age
* HbA1c ≥ 58 mmol/mol
* Currently using CGM or FGM
* To have a possibility to download and share FGM/CGM data

Exclusion Criteria:

* Type 2 diabetes
* Diabetes duration <1 year
* Long-term Systemic glucocorticoid treatment during the last 3 months
* Planned or changed treatment the last 3 months regarding MDI vs. Insulin pump or added or stopped CGM or FGM therapy
* Current or planned pregnancy or breastfeeding during the next 12 months
* Planned move during the next 12 months making it not possible to participate in study activities
* Other reason determined by the investigator not being appropriate for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to 18 weeks
  Change in HbA1c from baseline to week 18

SECONDARY OUTCOMES:
Time in Range | from baseline to 18 weeks
  Change in Time in Range (4-10mmol/l) and from Baseline to week 18
Mean glucose levels | from baseline to 18 weeks
  Change in mean glucose levels from baseline to 18
Time above range | from baseline to 18 weeks
  Change in time above range (glucose values above 10mmol/L) from baseline to 18 weeks
HbA1c at week 32 | From baseline to 18 weeks
  Change in HbA1c from baseline to week 32
HbA1c at week 52 | From baseline to 52 weeks
  Change in HbA1c from baseline to week 52

OTHER OUTCOMES:
Mean Glucose at week 32 and 52 | From baseline to 32 and 52 weeks
  Change in mean glucose from baseline to week 32 and 52
Time below range week 18, 32 and 52 | From baseline to 18, 32 and 52 weeks
  Change in time below range (glucose values below 4.0mmol/l) from baseline to week 18, 32 and 52
Time above range weeks 32 and 52 | From baseline to weeks 32 and 52
  Change in time above range from baseline to 32 and 52 weeks
Glycaemic variability - Standard deviation | From baseline to weeks 18, 32 and 52
  Change in glycaemic variability from baseline to 18, 32 and 52 weeks using Standard deviation
Glycaemic variability - Coefficient of variation | From baseline to weeks 18, 32 and 52
  Change in glycaemic variability from baseline to 18, 32 and 52 weeks using Coefficient of variation
Glycaemic variability - Mage | From baseline to weeks 18, 32 and 52
  Change in glycaemic variability from baseline to 18, 32 and 52 weeks using MAGE
DTSQ | From baseline to weeks 18, 32 and 52
  Change in Diabetes Treatment and satisfaction (DTSQ) score from baseline to 18, 32 and 52 weeks. DDS is a 6 pt Lickert scale with 28 questions
Hypoglycaemic confidence | From baseline to weeks 18, 32 and 52
  Change in Hypoglycaemic confidence score from baseline to 18 and 52 weeks. The hypoglycemic confidence scale is a 4pt Lickert scale with 9 questions
Diabetes distress scale | From baseline to weeks 18, 32 and 52
  Change in Diabetes distress score (DDS) score from baseline to 18 and 52 weeks. DDS is a 6 pt Lickert scale with 28 questions

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Hosptial Group, Uddevalla, Sweden

REFERENCES:
- [Derived] Olafsdottir AF, Sveen KA, Wijkman M, Hallstrom S, Nilsson PH, Sterner Isaksson S, Holmer H, Ekstrom M, Imberg H, Lind M. Systematic intensive therapy in addition to continuous glucose monitoring in adults with type 1 diabetes: a multicentre, open-label, randomised controlled trial. Lancet Reg Health Eur. 2025 Oct 16;59:101485. doi: 10.1016/j.lanepe.2025.101485. eCollection 2025 Dec. PMID 41142656
- [Derived] Olafsdottir AF, Lind M. Evaluating a systematic intensive therapy using continuous glucose monitoring and intermittent scanning glucose monitoring in clinical diabetes care: a protocol for a multi-center randomized clinical trial. Front Clin Diabetes Healthc. 2023 Oct 18;4:1247616. doi: 10.3389/fcdhc.2023.1247616. eCollection 2023. PMID 37920192